CLINICAL TRIAL: NCT01286025
Title: A Randomized Crossover Study to Compare the Critical Thinking of Medical Students When Using Video-based or Written Cases
Brief Title: Comparing the Effect of Video-cases and Text-cases on Medical Students' Learning in Tutorial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Responsible Party: Graham T. McMahon MD MMSc, Harvard Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: M15700-101
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Education, Medical; Education, Medical, Undergraduate; Problem-based Learning; Problem Solving; Interactive Tutorial
Keywords: medical education; problem-based learning; interactive tutorial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video modality (Active Comparator)
  Interventions: Behavioral: video case modality
- Text modality (Active Comparator)
  Interventions: Behavioral: Text case modality

INTERVENTIONS:
Behavioral: video case modality — Patients whose case histories are pathophysiologically illustrative will be recruited, and interviewed on video. Their stories will be edited and divided into sections, and combined with the patient's laboratory, imaging, and pathological reports when appropriate
  Arms: Video modality
Behavioral: Text case modality — Patients whose case histories are pathophysiologically illustrative will be recruited, and interviewed on video. Their stories will be edited and divided into sections, and combined with the patient's laboratory, imaging, and pathological reports when appropriate. The transcript of these video-recordings will form the basis of the text-based case presentation modality.
  Arms: Text modality

SUMMARY:
This study is designed to examine how the type of learning case affects the thinking of medical students in tutorial

DETAILED DESCRIPTION:
Tutorials at Harvard Medical School use problem-based learning with written cases. Students work in groups under the supervision of a tutor who guides their exploration of the material. As students progress through the curriculum there is an opportunity to advance the complexity of the material they are presented with. Video-based patient case studies have been shown to improve critical thinking ratios in paediatric medical student problem-based learning exercises, and time spent on data exploration, theory building and theory evaluation in postgraduate residency programs. We hypothesize that video provides a stimulus that improves cognitive processing and critical thinking among medical students, as compared to working from the text-based transcript of the same case.

ELIGIBILITY:
Inclusion Criteria:

* medical student participating in the endocrine and reproductive pathophysiology course at Harvard Medical School

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Overall ratio of deep to superficial thinking | Four 90-minute tutorial sessions
  Depth of thinking will be evaluated using the method of Kamin et al. Transcription of each tutorial will be divided into utterances. Each utterance will be coded for depth of thinking (deep vs. superficial). The ratio of deep to superficial thinking by case modality will be reported.

SECONDARY OUTCOMES:
Distribution of learning activities | Four 90-min tutorial sessions
  Transcription of each tutorial will be divided into utterances. Each utterance will be coded by learning domain (identification, description, exploration, integration, and application. The distribution of domains by case modality will be reported.
Preferences of students for each case modality | 5 weeks
  Students will be surveyed regarding their preferences for video- vs. text-based case presentation modality using a Likert-scale
Preferences of tutors for each case modality | 5 weeks
  Tutors will be surveyed regarding their preferences for video- vs. text-based case presentation modality using a Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Graham T McMahon, MD MMSc, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States